CLINICAL TRIAL: NCT01598909
Title: Efficacy of Arnica D1 Ointment After Upper Blepharoplasty: a Randomized, Double-blind Placebo-controlled Study
Brief Title: Efficacy of Arnica D1 Ointment After Upper Blepharoplasty
Acronym: ARINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wynand BWH Melenhorst, MD (Other)
Responsible Party: Sponsor-Investigator, Wynand BWH Melenhorst, MD, MD, PhD, Isala
Organization: Isala (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARINE Study
Record Dates: First submitted 2012-05-12; First posted 2012-05-15 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Blepharoplasty; Upper Eyelid Blepharoplasty
Keywords: blepharoplasty; arnica; homeopathy
MeSH Terms: interventions — Arnicae flos extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arnica ointment (Active Comparator)
  Interventions: Drug: Arnica
- Placebo ointment (Placebo Comparator)
  Interventions: Drug: Placebo ointment
- Control (No Intervention)

INTERVENTIONS:
Drug: Arnica — Application of Arnica ointment periorbitally
  Arms: Arnica ointment
Drug: Placebo ointment — Application of Arnica ointment, twice a day, for the period of one week.
  Arms: Placebo ointment

SUMMARY:
Arnica ointment is currently used in homeopathic preparations for strains and bruises. In the field of plastic surgery, some surgeons advise patients undergoing blepharoplasty to use Arnica in order to prevent postoperative ecchymosis, swelling and pain. Thus far, no decent study evaluated the efficacy of topical Arnica ointment in reducing ecchymosis or surgical outcome after upper blepharoplasty. We hypothesize that application of Arnica ointment postoperatively will reduce the development of ecchymosis and improve outcome.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing primary blepharoplasty

Exclusion Criteria:

* use of anticoagulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Surgical outcome | 7 days and 6 weeks postoperatively
  Overall judgment of surgical outcome, based on the combined analysis of the amount of ecchymosis, swelling and redness, by an unrelated, uninvolved and "blinded" plastic surgeon.

SECONDARY OUTCOMES:
amount of tissue swelling; redness; pain; postoperative recovery; patient satisfaction | 3, 7 and 42 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: W Melenhorst, MD PhD, Principal Investigator — Isala
Locations (1):
- Isala Klinieken, Zwolle, Netherlands